CLINICAL TRIAL: NCT07318363
Title: IGNITE-TX Phase III: (Identifying Individuals for Genetic Testing & Treatment) Intervention
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-1276; NCI-2025-09245 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-12-29; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Communication; Informed Decision-making
MeSH Terms: conditions — Communication | interventions — Genetic Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of Care (Experimental): ARRs: No active efforts will be made to ensure that ARRs complete genetic testing or to support family communication and education during the period in which primary study outcomes are being evaluated.
  Interventions: Other: IGNITE-TX program; Other: Genetic Counseling and Testing
- Free Genetic Counseling and Testing (Experimental): ARRs: A letter will be provided to the ARR with instructions on how to access genetic counseling and free testing through a telegenetics company (Appendix E).
  Interventions: Other: IGNITE-TX program; Other: Genetic Counseling and Testing
- IGNITE-TX Intervention (Experimental): ARRs: The relatives will receive instructions with a code to access the IGNITE-TX Hub (Appendix K & L). Family Genetic Navigators will support this process by reaching out and guiding relatives through the process.
  Interventions: Other: IGNITE-TX program; Other: Genetic Counseling and Testing
- IGNITE-TX Intervention + Free Genetic Counseling and Testing (Experimental): ARRs: The relative will be sent instructions to access free counseling and testing, as well as a unique code to log into the IGNITE-TX Hub (Appendix K & L). Family Genetic Navigators will support this process by reaching out and guiding relatives through both resources.
  Interventions: Other: IGNITE-TX program; Other: Genetic Counseling and Testing

INTERVENTIONS:
Other: IGNITE-TX program — Participants will complete a questionnaire
Other: Genetic Counseling and Testing — Participants will complete a questionnaire

SUMMARY:
This trial aims to implement and compare an evidence- and theory-based intervention strategy (IGNITE-TX Intervention) to support probands and their ARRs in family communication, informed decision-making, and navigation to CGT with standard of care, free genetic testing/counseling, and intervention with free genetic testing/counseling.

DETAILED DESCRIPTION:
Primary Objectives:

1. Determine the impact of IGNITE-TX on the uptake of cascade genetic testing (CGT) in at-risk relatives (ARRs) at 6 months.
2. Use a mixed methods approach, guided by the NIMHD framework, to evaluate the impact of IGNITE-TX on informational, social, and emotional support outcomes within families at 6 months.
3. Employ formative and process evaluations and stakeholder engagement to guide IGNITE-TX implementation and dissemination through the RE-AIM QuEST framework.

Secondary Objective:

1. Analyze the correlation of CGT completion rates within families to understand the influence of familial relationships on genetic testing uptake.

Exploratory Objective:

Evaluate the effectiveness of social media as a mechanism to drive outreach, recruitment, and engagement with the IGNITE-TX intervention.

ELIGIBILITY:
Inclusion Criteria:

Probands:

1. 18 years of age or older
2. Speaks and reads English or Spanish
3. Resides in the United States
4. Has a pathogenic or suspected pathogenic variant in BRCA1, BRCA2, MLH1, MSH2/EPCAM, MSH6, or PMS2*
5. Has access to the internet or phone and can send and receive email and/or text messages at a US telephone number.
6. Attests to have at least one at-risk relative who meets inclusion criteria for first-degree relative *For cancer patients who are unaware of their mutation status, we will share existing local and national genetics resources, like those provided in the usual care family letter.

At-Risk Relatives (ARR):

1. 18 years of age or older
2. Speaks and reads English or Spanish
3. Resides in the United States
4. Has a first or second degree relative who has a deleterious/suspected deleterious HBOC or LS variant present
5. Has access to internet or phone and can send and receive email and/or text messages at a US telephone number

Exclusion Criteria:

Probands:

1. Has no eligible at-risk relatives (ARRs) or is unable/unwilling to provide their contact information
2. Has negative germline genetic testing or only variant of uncertain significance
3. Unwilling or unable to provide consent

At-Risk Relatives (ARR):

1. Unwilling or unable to provide consent
2. Reports no known HBOC or LS variant within the family
3. Has already been tested for the variant identified in the proband
4. Already listed as an ARR for another proband

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jose Alejandro Rauh-Hain, MD, MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org